CLINICAL TRIAL: NCT07338240
Title: Real-Time Validation and Feasibility of the SOFA-2 Score in Adult Intensive Care Units in Türkiye (TR-SOFA2): A Multicenter Prospective Observational Study
Brief Title: SOFA-2 Score in Turkish ICUs
Acronym: TR-SOFA2
Status: Recruiting | Type: Observational
Sponsor: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Cenk Kirakli, M.D., Professor, Intensive Care Unit, Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital
Other Study IDs: IGHCEAH-ICU-8
Record Dates: First submitted 2025-12-22; First posted 2026-01-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Intensive Care Unit Patients; Critically Ill Intensive Care Unit Patients
Keywords: SOFA-2 Score; Critical Illness; ICU Mortality; Prognostic Scoring System
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult ICU Patients: This cohort consists of adult patients aged 18 years or older who are admitted to participating intensive care units in Türkiye and remain in the ICU for more than 24 hours. Patients are enrolled prospectively and followed from ICU admission until ICU discharge or death. Clinical and laboratory data routinely collected during standard care are used to calculate SOFA and SOFA-2 scores. No study-specific interventions, additional diagnostic procedures, or changes to standard clinical

SUMMARY:
This study aims to evaluate how well a new scoring system called the Sequential Organ Failure Assessment-2 (SOFA-2) works in adult intensive care units in Türkiye.

SOFA-2 is designed to measure the severity of organ dysfunction in critically ill patients using routinely collected clinical and laboratory data. It is an updated version of the original SOFA score and reflects modern intensive care practices.

In this multicenter observational study, adult patients admitted to participating intensive care units will be followed during their ICU stay. SOFA and SOFA-2 scores will be calculated during the first 24 hours of admission, and in patients with longer stays, additional scores will be recorded. No additional tests or treatments will be performed as part of the study.

The main goal of the study is to examine the relationship between SOFA-2 scores and intensive care unit mortality. The results are expected to help clinicians better assess disease severity and outcomes in critically ill patients.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational study designed to evaluate the feasibility and prognostic performance of the Sequential Organ Failure Assessment-2 (SOFA-2) score in adult intensive care units across Türkiye.

Adult patients aged 18 years or older who are admitted to participating intensive care units and remain in the ICU for more than 24 hours will be eligible for inclusion. Pregnant patients, organ donors, patients younger than 18 years, and those with unknown ICU discharge outcomes will be excluded.

Demographic characteristics, reasons for ICU admission, comorbid conditions, and routinely collected clinical and laboratory data will be prospectively recorded using standardized case report forms. SOFA and SOFA-2 scores will be calculated based on data obtained during the first 24 hours following ICU admission. For patients with an ICU stay longer than 72 hours, additional SOFA and SOFA-2 scores will be recorded at 72 hours.

Patients will be followed until ICU discharge or death. No study-specific interventions, additional diagnostic procedures, or changes to standard clinical management will be implemented as part of the study.

The study will assess the feasibility of real-time SOFA-2 score calculation, evaluate its association with ICU mortality, and compare its prognostic performance with the original SOFA score. Analyses will account for the multicenter structure of the study and variations across participating intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Admission to a participating intensive care unit in Türkiye
* Intensive care unit stay longer than 24 hours

Exclusion Criteria:

* Patients younger than 18 years
* Pregnant patients
* Organ donors
* Patients with unknown intensive care unit discharge outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients admitted to participating intensive care units across Türkiye. Eligible participants are critically ill adults who require intensive care monitoring and treatment and remain in the intensive care unit for more than 24 hours. The study includes a broad and heterogeneous ICU population reflecting routine clinical practice and does not target a specific dise
Sampling Method: Non-Probability Sample
Enrollment: 5200 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Association Between 24-Hour SOFA-2 Score and ICU Mortality | 60 days after ICU admission
  The association between the total SOFA-2 score calculated within the first 24 hours of intensive care unit admission and all-cause ICU mortality. Higher scores show worse outcomes.

SECONDARY OUTCOMES:
Reclassification Performance of SOFA-2 Compared With SOFA | 60 days after ICU admission
  Comparison of patient risk classification between SOFA and SOFA-2 scores with respect to ICU mortality.Higher scores show worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, İzmir School of Medicine, Dr. Suat Seren Chest Disease and Thoracic Surgery Training and Research Hospital, Intensive Care Unit, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data related to baseline demographics, ICU admission characteristics, SOFA and SOFA-2 scores, and ICU outcomes that underlie the results reported in the primary publication will be shared. No direct identifiers or protected health information will be included.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 6 months after publication Ending 5 years after publication
Access Criteria: Supporting information and de-identified individual participant data will be made available upon reasonable request. Requests will be reviewed by the study steering committee, and access will be granted following approval of a methodologically sound proposal and execution of a data use agreement.

REFERENCES:
- [Background] Ranzani OT, Singer M, Salluh JIF, Shankar-Hari M, Pilcher D, Berger-Estilita J, Coopersmith CM, Juffermans NP, Laffey J, Reinikainen M, Neto AS, Tavares M, Timsit JF, Arias Lopez MDP, Arulkumaran N, Aryal D, Azoulay E, Celi LA, Chaudhuri D, De Lange D, De Waele J, Dos Santos CC, Du B, Einav S, Engelbrecht T, Fazla F, Ferrer R, Finazzi S, Fujii T, Gershengorn HB, Greene JD, Haniffa R, Hao S, Hasan MS, Hollenberg S, Ippolito M, Jung C, Kirov M, Kobari S, Lakbar I, Lipman J, Liu V, Liu X, Lobo SM, Magatti D, Martin GS, Metnitz B, Metnitz P, Myatra SN, Oczkowski S, Paiva JA, Paruk F, Pekkarinen PT, Piquilloud L, Polkki A, Prescott HC, Blaser AR, Rezende E, Robba C, Rochwerg B, Ruckly S, Samei R, Schenck EJ, Secombe P, Sendagire C, Siaw-Frimpong M, Simpkin AJ, Soares M, Summers C, Szczeklik W, Takala J, Tanaka S, Tricella G, Vincent JL, Wendon J, Zampieri FG, Rhodes A, Moreno R. Development and Validation of the Sequential Organ Failure Assessment (SOFA)-2 Score. JAMA. 2025 Dec 16;334(23):2090-2103. doi: 10.1001/jama.2025.20516. PMID 41159833
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069